CLINICAL TRIAL: NCT02216708
Title: Comparison of Rapid and Slow Rehydration of Severely Malnourished Children Suffering From Dehydrating Diarrhoea and Impact on Renal Function and Subsequent Growth of Children
Brief Title: Slow Versus Rapid Rehydration of Severely Malnourished Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-11004
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2011-03

CONDITIONS: Diarrhea
Keywords: Severe malnutrition; severe dehydration; cholera
MeSH Terms: conditions — Diarrhea; Malnutrition; Dehydration; Cholera

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intravenous fluid for rehydration rapidly over 6 hours (Experimental): intravenous fluid for rehydration rapidly over 6 hours
  Interventions: Other: Rapid dehydration
- receive slow rehydration recommended by WHO (12 hours) (Experimental): receive intravenous fluid followed by ORS (slow rehydration recommended by WHO) over 12 hours
  Interventions: Other: Slow rehydration

INTERVENTIONS:
Other: Rapid dehydration
  Arms: intravenous fluid for rehydration rapidly over 6 hours
Other: Slow rehydration
  Arms: receive slow rehydration recommended by WHO (12 hours)

SUMMARY:
The recommendation for correction of dehydration of severely malnourished children with diarrhoea includes oral rehydration and if parenteral rehydration is necessary (for example, in severe dehydration) to infuse intravenous fluids very slowly due to the concern of heart failure. There is not enough evidence to convince some of the physicians dealing with severely malnourished children with dehydrating diarrhoea (for example, cholera) that rapid rehydration per se is associated with increased incidence of over hydration and heart failure. And whether this approach is applicable in the management of severely malnourished children with severe cholera, which usually require rapid correction of water and electrolyte deficits for prevention of deaths due to hypovolaemic shock and other complications, has not been studied carefully. Recently, we have demonstrated that rapid intravenous rehydration (within 4 to 6 hours) of severely malnourished children with dehydrating cholera replacing appropriate amount of fluid was found to be safe. We feel that rapid rehydration would help in improving the renal function, acidosis and thus improve appetite and reduce ORS failure subsequently. Since our study was uncontrolled, so we have planned a randomised controlled study with adequate sample of 250 participants; 125 will be rehydrated slowly (over 10 to 12 hours) following WHO guideline and 125 patients will be rehydrated with intravenous fluid over 6 hours. Children of either gender, age 6 to 60 months, severely malnourished (Wt for length <-3 Z score of WHO growth chart or with nutritional oedema) with a history of watery of <24 hours with signs severe dehydration attending the ICDDRB Dhaka hospital will be asked to participate in this study. After the parents'/Legal guardian's consent, the children will be transferred to the study ward and will be treated according to the protocol. All children will receive similar treatment except the mode of rehydration, different for the two groups. The children will be closely monitored throughout the study period. The primary outcomes incidence of over hydration and ORS failure and secondary outcomes improvement of renal function and improvement of appetite measured by the food intake will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

1. History of acute watery diarrhoea of <24 hours.
2. Either sex.
3. Severe dehydration according to WHO guidelines
4. Wt for length/wt for age < -3 SD of WHO growth standard with or without oedema.(malnutrition)
5. Consent given by the parents or legal guardian

Exclusion Criteria:

1. Bloody diarrhoea.
2. Severe infection (e.g. severe pneumonia, clinical sepsis, septic shock, meningitis).
3. Those who received antibiotics/antimicrobial for the current illness

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Incidence of over- hydration | 7 days
Proportion of patient with ORS failure/ requirement of unscheduled IV therapy | 7 days

SECONDARY OUTCOMES:
Proportion of patient with acidosis and increased serum creatinine after 24 hours | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- icddr,b Dhaka Hospital, Dhaka, Bangladesh